CLINICAL TRIAL: NCT02636790
Title: Is Prioritization of the Sinus Surgical Waitlist Required?
Brief Title: Early Versus Late Surgical Wait Times
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Arif Janjua, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H15-02020
Record Dates: First submitted 2015-12-03; First posted 2015-12-22 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery wait time (< 8 weeks) (Active Comparator): Outcomes of patients with sinus surgery of less than 8 weeks.
  Interventions: Procedure: Surgery wait time
- Surgery wait time (> 1 year) (Active Comparator): Outcomes of patients with sinus surgery of more than 1 year.
  Interventions: Procedure: Surgery wait time

INTERVENTIONS:
Procedure: Surgery wait time — VCH CRS patients need a waitlist system that promotes wellness and ensures care that focuses on quality - this can be achieved with a prioritized waitlist based on quality of life improvement and decreased healthcare expenditure.

SUMMARY:
The sinus surgical wait list in British Columbia continues to grow. The current wait list is beyond what is acceptable by the province's standard; however, this is not likely to improve given the budget constraints of the health care system. The outcome of having patients to wait longer than medically reasonable for surgery, not only affects the patients' quality of life but presents financial difficulties, both directly to the patient, the healthcare system and the economy as a whole. Therefore, the investigators need to determine which patients need to be prioritized for surgery. The investigators will follow two groups of patients - one group from Stanford University who get surgery always before 8 weeks and compare them to patients on the VGH wait list which is often more than one year.

DETAILED DESCRIPTION:
Introduction Five percent of Canadians suffer from Chronic Rhinosinusitis (CRS) based on a national survey.1 CRS sufferers have debilitating facial pain, nasal congestion, nasal discharge and poor sense of smell. Relative to other chronic diseases, the quality of life of patients suffering with CRS is comparable to diseases such as congestive heart failure, chronic obstructive pulmonary disease, angina and back pain.3 Currently, CRS patients in Vancouver, British Columbia wait just over a year for surgery. British Columbia's (BC) health care policy recommends that CRS patients waiting for surgery be done in twelve weeks. It is well recognized that patients who wait longer than medically reasonable for surgery result in an excess costs, both directly to the patient, the healthcare system and the economy as a whole.5 Unfortunately, no studies done in Canada have illustrated the direct and indirect costs associated with CRS annually.

Patients' waiting time for elective sinus surgery in BC has come under public scrutiny in recent years. As a result, policy-makers are keen to address this waitlist issue.4 The government has identified sinus surgery as an elective day procedure that requires the Patient Focused Fund (PFF) to increase volume and address its disproportionately large waitlist. This likely has resulted in savings to VCH patients and the BC Health Ministry that would not have occurred had the PFF not been initiated. However, policy-makers must explore other innovate ways to supplement the PFF to provide further savings to VCH patients and the BC health care system.

An approach that has been adopted by other specialities such as orthopaedics, ophthalmology, and radiology is the use of a validated tool to prioritize waitlists.6-8 There are no validated tools published for prioritizing sinus surgery waitlists. The Canadian Institutes of Health Research provided funding to establish the Western Canada Waiting List Project (WCWL) to "improve the fairness of the health care system so that Canadians' access to appropriate and effective medical services is prioritized on the basis of need and potential benefit."9 Despite the work done by the WCWL being limited to five clinical areas (cataract surgery; general surgery procedures; hip and knee replacement; magnetic resonance imaging (MRI) scanning, and children's mental health), the methodology utilized in establishing their prioritization tool can be used to establish one for the sinus surgery waitlist;10 The impact of chronic diseases, including CRS, varies among patients11; therefore, prioritizing patients based on clinical measurements and cost-effectiveness from an individual and healthcare system perspective would be a novel approach to addressing waitlists for sinus surgery. Currently, VCH CRS patients are treated on a first come, first served basis. Despite this being the most transparent way of ordering the waitlist, the investigators feel VCH CRS patients need a waitlist system that promotes wellness and ensures care that focuses on quality - this can be achieved with a prioritized waitlist based on quality of life improvement and decreased healthcare expenditure.

Prior to establishing a validated tool for the prioritization of sinus surgery waitlists, one must first determine if VCH patients and the BC health care system would benefit from prioritized surgery. Providing a solution to this question requires moderate amount of resources and would take several of years to complete. The investigators propose a feasibility study coupled with an economic evaluation to determine if the disproportionately long wait list faced by CRS patients can be optimized and thus improve patient outcomes.

Current State of Knowledge Researchers must determine if CRS patients and the BC health care system would benefit from a prioritized waitlist for sinus surgery. It is accepted that sinus surgery compared to medical therapy improves the quality of life of CRS patients.12-14 However, to determine whether VCH CRS patients would benefit from a prioritized waitlist, the investigators must answer the following questions. If patients were to have surgery sooner: 1) how does their quality of life change with time compared to those on the waitlist? 2) do they experience a reduction in out of pocket costs?; 3) does the healthcare system experience a decrease in healthcare expenditure? and 4) is there are a subgroup of patients who would particularly benefit more than others from early surgical intervention? Providing this information is vital in determining if a prioritized waitlist would be beneficial for sinus surgery.

Patient Recruitment:

Recruitment of patients will occur at two centres. Patients classified as "prioritized surgery" will be recruited from Stanford Sinus Centre, Palo Alto, California. Patients classified as "standard waitlist" patients will be recruited from Vancouver General Hospital, Vancouver, Canada. The PI will identify consecutive patients that fit the inclusion/exclusion criteria and are being enrolled for sinus surgery. The study coordinator (or designate) will discuss the study with the identified patients and allow patients up to 7 days to provide consent.

On the day of consent:

A diagnosis of the patient's medical health will be conducted by the study investigators and a Lund-Mackay and Lund-Kennedy score systems will be used to assess the patient's chronic rhinosinusitis. Additionally, the state of the rhinosinusitis will be evaluated on the day of consent and on every subsequent follow-up visit. A questionnaire relating to demographics will be obtained as well (Appendix D).

Approach to Each Aim:

Aim 1: The investigators will compare how the quality of life of CRS patients change with time when prioritized to early surgical intervention compared to those on the standard waitlist.

All CRS patients participating in the study will fill in a disease-specific health related quality of life instrument for CRS patients known as the Sinonasal Outcome Test (SNOT-22) and two generic assessment of health status known as the WPAI-SHP and EQ-5D (Appendix A) every 2 months for 1 year.

The study coordinator (or designate) will contact patients every 2 months via email and provide them with a secure link to fill in each questionnaire. When questionnaires are complete, they will be saved directly into their medical records.

Rationale for Questionnaires: The Sinonasal Outcome Test (SNOT-22) is a validated questionnaire.16 SNOT-22 is a disease-specific health-related quality of life instrument in CRS patients. The EQ-5D has 5 questions addressing: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The Work Productivity and Activity - Specific Health Problem (WPAI:SHP) is a validated instrument to evaluate impairment of daily activities and work productivity associated with a specific health problem (Chronic Rhinosinusitis). The work productivity impairment domain is a sum of impairment in work productivity due to absenteeism and due to decreased productivity while working (presenteeism); this domain is assessed only in employed patients. The activity impairment domain is assessed in all participants regardless of their employment status and represents impairment in daily activities other than work.18 The investigators would prefer to use an easy to administer generic health measure like the EQ-5D compared to the WPAI-SHP, but during the feasibility stage, the investigators will administer both questionnaires and at the completion of the study determine the most appropriate questionnaire for this study.

Aim 2: To determine if patients prioritized to early surgical intervention experience a reduction in out of pocket costs compared to patients on the standard waitlist.

All CRS patients participating in the study will fill in a questionnaire regarding personal costs incurred over 1 year. To ensure the most accurate costs are tabulated, patients will fill in this questionnaire every two months (Appendix B).

The study coordinator (or designate) will contact patients every two months via email and provide them with a secure link to fill in questions from Appendix B similar to Aim 1. The study coordinator (or designate) will follow the same protocol of contacting the patient if the questionnaire is not filled in a timely manner. Patients can also complete this Aim on a hard copy similar to Aim 1.

To ensure the investigators were inclusive of all the cost incurred by CRS patients, a sample population of 30 VCH CRS patients were surveyed. Moreover, a panel that included multiple Rhinologists and a Health Economist established questions that were pertinent to costs incurred by the patient that may have been overlooked by the sample population. This process ensures that the most accurate estimate of personal costs incurred by CRS patients while waiting for surgery and those prioritized to early surgery. (Appendix B) Aim 3: The investigators will determine if the Canadian health care system experiences a decrease in healthcare expenditure if CRS patients are enlisted for early surgical intervention versus patients on the standard waitlist.

When VCH CRS patients are addressing Aim 2, they will also have additional questions that pertain to costs incurred by the health care system (Appendix B). The PI will fill in a questionnaire regarding costs incurred by the health care system for 1 year for each patient when there is a believed cost to the public system that is atypical compared with expected costs (Appendix C). During each clinical for each patient, the PI will tabulate the costs incurred during the patient's clinical visit.

Like in Aim 2, a panel consisting of multiple Rhinologists established Appendix C. Moreover, during three clinical days by the PI, extra costs incurred by the VCH health care system were noted and included into Appendix C.

Aim 4: The investigators will determine if there is a subgroup of CRS patients who would benefit from early surgical intervention.

Stratification of VCH CRS patients and determining if patients benefited from early surgical intervention will be established through demographic information, clinical findings and comparison of outcomes obtained in Aims 1-3. Demographic information will be obtained on the day consent is obtained (Appendix D). The PI will also complete a standardized consultation/follow-up form for each visit to report clinical findings.

The PI will also complete a standardized consultation/follow-up form, including an evaluation of healing subsequent to nasal surgery based on the Lund-Kennedy score, for each visit to document clinical findings.

Analysis:

Pre-Study Sample Size Calculation - Sample size for comparison on average difference in SNOT-22 scores between two equally sized group over time followed the Diggle et al formula.19 Based on an effect size of 9 points15 between the early intervention and standard waitlist patients, type 1 probability of 5% (α = 0.05), a type 2 probability of 20% (β = 0.20), standard deviation of 20 from pre- and post surgical values15 and 6 measurements of SNOT-22 over 12 months, the assumed correlation (p) will range from 0.75 and 1.00 if 124 to 156 patients are recruited, therefore allowing for a conservative estimate of 10% drop-out.

Post-Study Completion - Aim 1 will be analyzed using 2-sample t-test. The investigators will conduct a cost-utility analysis to evaluate Aims 2 and 3. the investigators assume the cost of surgery for the early intervention group will be the same as those who will receive in it on the standard waitlist; therefore, this cost will be removed from the early intervention group. The economic model will evaluate costs and utilities (measured by EQ-5D and WPAI-SHP) and calculate incremental cost-effectiveness ratios (ICERs). The time horizon for this evaluation will be 1 year. No other discounting of costs or utilities is required given this time horizon. Uncertainty around the ICERs will be quantified using bootstrapping. Aim 4 will be analyzed using linear regression models. The best-fit model will provide insight to sub-population of CRS patients who would benefit from early surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CRS based on 2 major symptoms (congestion, facial pain, nasal obstruction, nasal discharge, decreased sense of smell) and evidence of sino-nasal inflammation on CT scan and nasal endoscopy. Symptoms must also be present for >12 weeks.

Exclusion Criteria:

* History of or requiring surgery for a sino-nasal tumour

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Questionnaire relating to demographics. | 30 min to complete questionnaire (once)
  Patient demographic information to be completed once after surgery to determine if there is a distinct group of chronic Rhinosinusitis patients who would benefit from early surgical intervention.
Change relating to personal costs over 1 year following surgery. | 30 min to complete questionnaire, every two months for 1 year (post-surgery).
  Personal costs related to surgical wait times.
Change to the quality of life over 1 year following surgery based on the WPAI-SHP questionnaire. | 10 min to complete questionnaire, every two months for 1 year (post-surgery).
  The questionnaire WPAI-SHP relates to quality of life after surgery. The Work Productivity and Activity - Specific Health Problem (WPAI:SHP) is a validated instrument to evaluate impairment of daily activities and work productivity associated with a specific health problem (Chronic Rhinosinusitis).
Change to the quality of life over 1 year following surgery based on the SNOT-22 questionnaire. | 10 min to complete questionnaire, every two months for 1 year (post-surgery).
  The questionnaire SNOT-22 relates to quality of life after surgery. SNOT-22 is a disease-specific health-related quality of life instrument in CRS patients.
Change to the quality of life over 1 year following surgery based on the EQ5-D questionnaire. | 10 min to complete questionnaire, every two months for 1 year (post-surgery).
  The questionnaire EQ5-D relates to quality of life after surgery. The EQ-5D has 5 questions addressing: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Arif Janjua, MD, Principal Investigator — UBC
Locations (2):
- Canada (2):
  - UBC - Department of Surgery Division of Otolaryngology - Head and Neck Surgery, Vancouver, British Columbia
  - UBC, Vancouver, British Columbia

REFERENCES:
- [Background] Chen Y, Dales R, Lin M. The epidemiology of chronic rhinosinusitis in Canadians. Laryngoscope. 2003 Jul;113(7):1199-205. doi: 10.1097/00005537-200307000-00016. PMID 12838019
- [Background] Cherry DK, Woodwell DA. National Ambulatory Medical Care Survey: 2000 summary. Adv Data. 2002 Jun 5;(328):1-32. PMID 12661586
- [Background] Gliklich RE, Metson R. The health impact of chronic sinusitis in patients seeking otolaryngologic care. Otolaryngol Head Neck Surg. 1995 Jul;113(1):104-9. doi: 10.1016/S0194-59989570152-4. PMID 7603703
- [Background] Mickleburgh, R. (2013, January 18). Ministers says BC wait lists too long. The Globe and Mail, Health Care, http://m.theglobeandmail.com/news/british-columbia/minister-says-bc-wait-lists-too-long/article7508904/?service=mobile (accessed on January 30, 2013).
- [Background] The economic cost of wait times in Canada. Retrieved from www.cma.ca/multimedia/CMA/Content.../EconomicReport.pdf (accessed on February 2, 2013).
- [Background] Conner-Spady BL, Sanmugasunderam S, Courtright P, Mildon D, McGurran JJ, Noseworthy TW; Steering Committee of the Western Canada Waiting List Project. The prioritization of patients on waiting lists for cataract surgery: validation of the Western Canada waiting list project cataract priority criteria tool. Ophthalmic Epidemiol. 2005 Apr;12(2):81-90. doi: 10.1080/09286580590932770. PMID 16019691
- [Background] Conner-Spady B, Estey A, Arnett G, Ness K, McGurran J, Bear R, Noseworthy T; Steering Committee of the Western Canada Waiting List Project. Prioritization of patients on waiting lists for hip and knee replacement: validation of a priority criteria tool. Int J Technol Assess Health Care. 2004 Fall;20(4):509-15. doi: 10.1017/s0266462304001436. PMID 15609803
- [Background] Hadorn DC; Steering Committee of the Western Canada Waiting List Project. Developing priority criteria for magnetic resonance imaging: results from the Western Canada Waiting List Project. Can Assoc Radiol J. 2002 Oct;53(4):210-8. PMID 12391927
- [Background] Noseworthy TW, McGurran JJ, Hadorn DC; Steering Committee of the Western Canada Waiting List Project. Waiting for scheduled services in Canada: development of priority-setting scoring systems. J Eval Clin Pract. 2003 Feb;9(1):23-31. doi: 10.1046/j.1365-2753.2003.00377.x. PMID 12558699
- [Background] Ben-Shlomo Y, Kuh D. A life course approach to chronic disease epidemiology: conceptual models, empirical challenges and interdisciplinary perspectives. Int J Epidemiol. 2002 Apr;31(2):285-93. No abstract available. PMID 11980781
- [Background] Western Canada Waiting List Investigators .(2013). Retrieved on February 2, 2013 from http://www.wcwl.ca/.
- [Background] Damm M, Quante G, Jungehuelsing M, Stennert E. Impact of functional endoscopic sinus surgery on symptoms and quality of life in chronic rhinosinusitis. Laryngoscope. 2002 Feb;112(2):310-5. doi: 10.1097/00005537-200202000-00020. PMID 11889389
- [Background] Smith TL, Kern R, Palmer JN, Schlosser R, Chandra RK, Chiu AG, Conley D, Mace JC, Fu RF, Stankiewicz J. Medical therapy vs surgery for chronic rhinosinusitis: a prospective, multi-institutional study with 1-year follow-up. Int Forum Allergy Rhinol. 2013 Jan;3(1):4-9. doi: 10.1002/alr.21065. Epub 2012 Jun 26. PMID 22736422
- [Background] Smith TL, Mendolia-Loffredo S, Loehrl TA, Sparapani R, Laud PW, Nattinger AB. Predictive factors and outcomes in endoscopic sinus surgery for chronic rhinosinusitis. Laryngoscope. 2005 Dec;115(12):2199-205. doi: 10.1097/01.mlg.0000182825.82910.80. PMID 16369166
- [Background] Bhattacharyya N, Orlandi RR, Grebner J, Martinson M. Cost burden of chronic rhinosinusitis: a claims-based study. Otolaryngol Head Neck Surg. 2011 Mar;144(3):440-5. doi: 10.1177/0194599810391852. Epub 2011 Feb 3. PMID 21493210
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277
- [Background] EuroQoL Group. EQ-5D. [Online] [Cited: January 30, 2013.] http://www.euroqol.org/.
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Diggle, P.J., Heagerty, P., Liang K-Y. and Zeger, S.L. (2002). Analysis of Longitudinal Data (second edition). Oxford: Oxford University Press.